CLINICAL TRIAL: NCT05784441
Title: A Phase 1b Multicenter, Open-Label, Study of JNJ-90009530, an Autologous Anti-CD20 CAR-T Cell Therapy in Adult Participants With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study of JNJ-90009530 in Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma (r/r B-NHL)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90009530LYM1001; 90009530LYM1001 (Other: Janssen Research & Development, LLC); 2023-506259-97-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-03-03; First posted 2023-03-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory B Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-90009530 (Experimental)
  Interventions: Drug: JNJ-90009530

INTERVENTIONS:
Drug: JNJ-90009530 — JNJ-90009530, an autologous Chimeric Antigen Receptor (CAR) - T therapy targeting CD20
  Other Names: C-CAR066

SUMMARY:
The goal of this multicenter study is to test JNJ-90009530 in Relapsed or Refractory Non-Hodgkin Lymphoma Patients. The main questions the study aims to answer are:

* can a dose of JNJ-90009530 be determined that is safe and well tolerated by patients.
* will JNJ-90009530 help patients achieve a response and for how long?

ELIGIBILITY:
Key Inclusion Criteria

* Participant must be greater than or equal to (>=) 18 years of age, at the time of signing informed consent
* All participants must have relapsed or refractory disease for each histologic subtype

  * Mature aggressive large B cell NHL and Follicular Lymphoma Grade 3b: Participants must have >= 2 lines of systemic therapy or >=1 line of systemic therapy in case of participants ineligible for high-dose chemotherapy and autologous Hematopoietic stem cell transplantation (HSCT). Participants also must have had exposure to an anthracycline and an anti-CD20 targeted agent
  * Follicular lymphoma Grade 1-3a and Marginal Zone Lymphoma: Participants must have >=2 prior lines of anti-neoplastic systemic therapy. Participants also must have prior exposure to an anti-CD20 monoclonal antibody
* Tumor must be cluster of differentiation (CD) 20 positive
* Measurable disease as defined by Lugano 2014 classification
* Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1

Key Exclusion Criteria

* Diagnosis of Human herpes virus (HHV) 8-positive Diffuse large B Cell lymphoma (DLBCL)
* Prior allogeneic Hematopoietic stem cell transplantation (HSCT)
* Autologous stem cell transplant within 12 weeks of chimeric antigen receptor (CAR) T cell infusion
* Uncontrolled active infections
* History of deep vein thrombosis or pulmonary embolism within six months of infusion (except for line associated deep vein thrombosis [DVT])
* History of stroke, unstable angina, myocardial infarction, congestive heart failure ( New York Heart Association [NYHA] Class III or IV), severe cardiomyopathy or ventricular arrhythmia requiring medication or mechanical control within 6 months of screening
* History of a seizure disorder, dementia, cerebellar disease or neurodegenerative disorder
* Known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system
* Active central nervous system (CNS) involvement by malignancy
* Current active liver or biliary disease (except for Gilbert's syndrome or asymptomatic gallstones)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2040-01-03 (Estimated)

PRIMARY OUTCOMES:
Calculate the Occurence of Adverse Events | up to 24 months
  The safety and tolerability will be measured by recording the occurence and severity of all adverse events or dose limiting toxicities that occur according to Common Terminology Criteria for Adverse Events (CTCAE) criteria version 5.0
Determine Recommended Phase 2 dose (RP2D) | up to 24 months
  Employ a Bayesian optimal interval (BOIN) design and determine the RP2D with review of the number of dose-limiting toxicities

SECONDARY OUTCOMES:
Determine the Overall Response (OR) | up to 24 months
  Record the number of subjects who have a complete response (CR) or partial response (PR) by radiographical assessment using Lugano Criteria 2014
Determine the time to response (TTR) | up to 24 months
  Record the number of days from the date of JNJ-90009530 infusion to a CR or PR
Determine the duration of response (DOR) | up to 24 months
  Record the number of days from the date of the first CR or PR to relapse or death.
Measure the amount of JNJ-90009530 in blood over time | up to 24 months
  Review pharmacokinetics (PK) of JNJ-90009530 by measuring the Chimeric Antigen Receptor (CAR) copy number over time by Quantitative polymerase chain reaction (qPCR).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (15):
- United States (7):
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Rutgers University, New Brunswick, New Jersey
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Medical Centre, Clayton
  - Austin Hospital, Heidelberg
  - Royal Brisbane and Women's Hospital, Herston
  - Westmead Hospital, Westmead
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency